CLINICAL TRIAL: NCT03578185
Title: Genomic Analysis to Identify a Predictive Biomarker for Immunotherapy
Acronym: LC_Biomarker
Status: Recruiting | Type: Observational
Sponsor: Se-Hoon Lee (Other)
Responsible Party: Sponsor-Investigator, Se-Hoon Lee, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Other Study IDs: Lung cancer Biomarker_2018
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The following analysis will be conducted using samples (tissue, blood, fecal material) form the patient who treated with immune checkpoint inhibitor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is designed to identify the predictive biomarker for immunotherapy using patient samples (tumor tissue, blood, fecal material) who treated with immune checkpoint inhibitor.

DETAILED DESCRIPTION:
[Sample acquisition]

* Informed consent is waived for those who agree to donate samples left over from other clinical trials or acquired for other purposes to be used for other research by the sign to master agreement in advance.
* The study will be conducted based on the purposes indicated in the master agreement signed by tissue donator [Clinical data acquisition]
* Baseline demographics: Sex, Birth date, expire date (last follow-up date for the survivals)
* Lung cancer treatment history: diagnosed date, treatment history (surgery, radiation therapy, chemotherapy, immunotherapy treatment history, and responses), general performance, metastatic sites
* Lung cancer histologic information: pathology, histologic subtype, EGFR mutation profile, ALK-rearrangement result

ELIGIBILITY:
Inclusion Criteria:

1. aged above or equal to 18
2. Histologically confirmed lung cancer patients
3. Patient treated with immune checkpoint inhibitor

Exculsion Criteria:

NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total of 800 lung cancer patients treated with immune checkpoint inhibitor Study will be initiated from the date of IRB approval to Dec. 2020 for those who signed for master agreement for tissue donation for research purposes.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
List of biomarkers | Baseline
  Neoantigen, tumor mutation burden, MHC compatibility, T-cell receptor and associated immune gene signature (IFN-r, interferons such as IL-2 and interleukin family), T-cell subset (T cell surface marker such as CD4+, CD7+, CD8+, CD16, CD34+, CD38+, CD56+, etc.), PD-1/PD-L1 expression, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Se-hoon Lee, MD, Study Chair — Samsung Medical Center
Locations (3):
- South Korea (3):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Seoul National University Hospital, Seoul, Joungro-gu
  - Asan Medical Center, Seoul, Songpa-gu

REFERENCES:
- [Background] Topalian SL, Weiner GJ, Pardoll DM. Cancer immunotherapy comes of age. J Clin Oncol. 2011 Dec 20;29(36):4828-36. doi: 10.1200/JCO.2011.38.0899. Epub 2011 Oct 31. PMID 22042955
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Brahmer JR, Drake CG, Wollner I, Powderly JD, Picus J, Sharfman WH, Stankevich E, Pons A, Salay TM, McMiller TL, Gilson MM, Wang C, Selby M, Taube JM, Anders R, Chen L, Korman AJ, Pardoll DM, Lowy I, Topalian SL. Phase I study of single-agent anti-programmed death-1 (MDX-1106) in refractory solid tumors: safety, clinical activity, pharmacodynamics, and immunologic correlates. J Clin Oncol. 2010 Jul 1;28(19):3167-75. doi: 10.1200/JCO.2009.26.7609. Epub 2010 Jun 1. PMID 20516446
- [Background] Patnaik A, Kang SP, Rasco D, Papadopoulos KP, Elassaiss-Schaap J, Beeram M, Drengler R, Chen C, Smith L, Espino G, Gergich K, Delgado L, Daud A, Lindia JA, Li XN, Pierce RH, Yearley JH, Wu D, Laterza O, Lehnert M, Iannone R, Tolcher AW. Phase I Study of Pembrolizumab (MK-3475; Anti-PD-1 Monoclonal Antibody) in Patients with Advanced Solid Tumors. Clin Cancer Res. 2015 Oct 1;21(19):4286-93. doi: 10.1158/1078-0432.CCR-14-2607. Epub 2015 May 14. PMID 25977344